CLINICAL TRIAL: NCT02545283
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase III Study of Idasanutlin, an MDM2 Antagonist, With Cytarabine Versus Cytarabine Plus Placebo in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study of Idasanutlin With Cytarabine Versus Cytarabine Plus Placebo in Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Acronym: MIRROS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped for futility based on efficacy results at the interim analysis; no unexpected safety findings were observed.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO29519; 2014-003065-15 (EudraCT Number)
Record Dates: First submitted 2015-08-31; First posted 2015-09-09 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; RG7388

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Idasanutlin plus Cytarabine (Experimental): Participants will receive induction therapy idasanutlin and cytarabine for 5 Days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or complete remission with incomplete blood count recovery (CRi), up to 28 additional days are allowed for blood count recovery, if needed.
  Interventions: Drug: Cytarabine; Drug: Idasanutlin
- Placebo plus Cytarabine (Placebo Comparator): Participants will receive induction therapy idasanutlin matching placebo and cytarabine for 5 days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin matching placebo and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or CRi, up to 28 additional days are allowed for blood count recovery, if needed.
  Interventions: Drug: Cytarabine; Other: Placebo

INTERVENTIONS:
Drug: Cytarabine — Participants will receive cytarabine 1 gram per square meter (g/m^2) intravenous (IV) infusion for 5 days of every treatment cycle.
Drug: Idasanutlin — Participants will receive idasanutlin 300 mg per oral (PO) twice daily (BID) (in Cycle 1) or once daily (QD) (in Cycles 2 and 3) for 5 days of every treatment cycle.
  Other Names: RG7388
  Arms: Idasanutlin plus Cytarabine
Other: Placebo — Participants will receive idasanutlin matching placebo PO BID or QD for 5 days of every treatment cycle.
  Arms: Placebo plus Cytarabine

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study designed to compare overall survival in participants with relapsed or refractory AML treated with idasanutlin in combination with cytarabine versus participants treated with placebo and cytarabine. Participants will receive induction treatment with idasanutlin/placebo and cytarabine (Cycle 1). Responding participants may continue to receive a maximum of further two cycles of consolidation (Cycle 2 and Cycle 3). Complete remission (CR), CR with incomplete platelet count recovery (CRp), overall remission rate (ORR), event-free survival (EFS) and percentage of participants with an allogeneic hematopoietic stem cell transplant (HSCT) will also be compared between treatment arms. This study will include participants with and without TP53 wild type (TP53 WT) mutations.

ELIGIBILITY:
Inclusion Criteria:

* Documented/confirmed first/second refractory/relapsed AML using World Health Organization classification, except acute promyelocytic leukemia
* No more than 2 prior induction regimens (excluding prior HSCT) in their first line treatment and one must have included cytarabine with an anthracycline (or anthracenedione)
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Adequate hepatic and renal function
* White blood cell (WBC) count at randomization less than or equal to (</=) 50000 cells per cubic millimeter (/mm^3)

Exclusion Criteria:

* First relapsed participants aged less than (<) 60 years with first CR duration greater than (>) 1 year
* Participants with prior documented antecedent hematological disorder (AHD)
* AML secondary to any prior chemotherapy unrelated to leukemia
* Participants who are either refractory to or relapsed within 90 days of receiving a regimen containing a cumulative dose of greater than or equal to (>/=) 18 g/m^2 of cytarabine
* Participants who have received allogeneic HSCT within 90 days prior to randomization
* Participants who have received immunosuppressive therapy for graft versus host disease or for engraftment syndrome after autologous stem cell transplantation within 2 weeks prior to randomization
* Prior treatment with an Murine Double Minute 2 (MDM2) antagonist
* Participants receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy within 30 days from first receipt of study drug
* Participants with a history of other malignancy within 5 years prior to screening except for malignancy that has been in remission without treatment for at least 2 years prior to randomization
* Participants who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Participants with extramedullary AML with no evidence of systemic involvement
* Pregnant or breastfeeding participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (7):
  - Northwell Health, Great Neck, New York
  - New York Medical College, Hawthorne, New York
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Abramson Cancer Center; Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - M.D. Anderson Cancer Center; Department of Hematology, Houston, Texas
- Australia (5):
  - Canberra Hospital; Haematology Department, Canberra, Australian Capital Territory
  - Concord Repatriation General Hospital; Haematology, Sydney, New South Wales
  - Royal Adelaide Hospital; Haematology Clinical Trials, Adelaide, South Australia
  - Geelong Hospital; Andrew Love Cancer Centre, Geelong, Victoria
  - Alfred Hospital; Clinical Haematology and Bone Marrow Transplantation, Melbourne, Victoria
- Lkh-Univ. Klinikum Graz; Klin. Abt. Für Hämatologie, Graz, Austria
- Belgium (3):
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - CHU Sart-Tilman, Liège
  - AZ Delta (Campus Rumbeke), Roeselare
- Juravinski Cancer Clinic; Clinical Trials Department, Hamilton, Ontario, Canada
- Finland (2):
  - Helsinki University Central Hospital; Hematology, Helsinki
  - Tampere University Hospital; Hematology, Tampere
- France (10):
  - Centre Hospitalier Uni Ire; Service Des Maladies Du Sang, Angers
  - Hopital Claude Huriez; Hematologie, Lille
  - Institut J Paoli I Calmettes; Onco Hematologie 2, Marseille
  - Hopital Hotel Dieu Et Hme;Hopital De Jour, Nantes
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - HOPITAL SAINT ANTOINE;Hematologie Clinique, Paris
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
  - IUCT Oncopole; Hematologie, Toulouse
  - Hopitaux De Brabois; Hematologie Medecine Interne, Vandœuvre-lès-Nancy
- Germany (9):
  - Uniklinik RWTH Aachen; Klinik IV; Klinik Hämatologie, Onkologie, Hämostaseologie und Stamm., Aachen
  - Universitätsklinikum Bonn; Med. Klinik und Poliklinik III; Hämatologie, Onkologie und Rheumatologie, Bonn
  - Klinikum Braunschweig; Medizinische Klinik III; Klinik für Hämatologie und Onkologie, Braunschweig
  - Klinikum Chemnitz gGmbH Krankenhaus Küchwald Klinik f.Innere Medizin III, Chemnitz
  - Klinik der Uni zu Köln; I. Med. Klinik, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik und Poliklinik I, Dresden
  - Medizinische Hochschule Hannover; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - Uni. der Johannes Gutenberg-Universitaet Mainz; III. Medizinische Klinik und Poliklinik, Mainz
  - Universitätsklinikum Marburg Zentrum f. Innere Medizin, Marburg
- Israel (4):
  - Shaare Zedek Medical Center; Hematology Dept., Jerusalem
  - Hadassah Ein Karem Hospital; Haematology, Jerusalem
  - Rabin Medical Center-Beilinson Campus;Hematology-Oncology, Petah Tikva
  - Ichilov Sourasky Medical Center; Heamatology, Tel Aviv
- Italy (14):
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - Az. Osp. S. Orsola Malpighi; Istituto Di Oncologia Seragnoli, Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST); Onco-Ematologia, Meldola, Emilia-Romagna
  - Az. Osp. S. Maria Delle Croci; U.O. Di Ematologia, Ravenna, Emilia-Romagna
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Oncologia; Clinica Ematologica, Udine, Friuli Venezia Giulia
  - Az. Osp. Uni Ria Policlinico Tor Vergata; Unita Di Ematologia, Rome, Lazio
  - IRCCS AOU S.Martino; Clinica Ematologica, Genoa, Liguria
  - ASST PAPA GIOVANNI XXIII; Ematologia, Bergamo, Lombardy
  - Ospedale San Raffaele, IRCCS, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - A.O. Universitaria San Luigi Gonzaga di Orbassano; Ambulatorio per le Malattie Rare del Polmone, Orbassano (TO), Piedmont
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
- Netherlands (2):
  - Academisch Medisch Centrum; Hematologie, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland, New Zealand
- Norway (2):
  - Haukeland Universitetssjukehus; Klinisk forskningspost, Bergen
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Complejo Hospitalario Arnulfo Arias Madrid; Servicio de Hematología, Panama City, Panama
- Russia (3):
  - "Hematological Scientific Center, Moscow
  - St. Petersburg State Medical University n.a. I.P. Pavlov; Hematology, transfusiology and transplanta, Saint Petersburg
  - FGBU "Federal Medical and Research Center named after V.A.Almazov" Russian Ministry of Health, Saint Petersburg
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- Switzerland (2):
  - Universitätsspital Basel; Hämatologie, Basel
  - Universitätsspital Zürich Medizin Hämatologie; Klinik für Hämatologie, Zurich
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - St Bartholomew's Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Montesinos P, Beckermann BM, Catalani O, Esteve J, Gamel K, Konopleva MY, Martinelli G, Monnet A, Papayannidis C, Park A, Recher C, Rodriguez-Veiga R, Rollig C, Vey N, Wei AH, Yoon SS, Fenaux P. MIRROS: a randomized, placebo-controlled, Phase III trial of cytarabine +/- idasanutlin in relapsed or refractory acute myeloid leukemia. Future Oncol. 2020 May;16(13):807-815. doi: 10.2217/fon-2020-0044. Epub 2020 Mar 13. PMID 32167393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 612 participants were screened, of which 447 patients were randomized as P53 tumor protein Wild Type (TP53 WT) population. TP53WT Population consists of mutation-defined Acute Myeloid Leukemia (AML) subpopulations FLT3, IDH2 and IDH1.
Groups:
- Placebo Plus Cytarabine: Participants received induction therapy idasanutlin matching placebo and cytarabine for 5 Days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin matching placebo and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or CRi, up to 28 additional days are allowed for blood count recovery, if needed.
- Idasanutlin Plus Cytarabine: Participants received induction therapy idasanutlin and cytarabine for 5 days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or complete remission with incomplete blood count recovery (CRi), up to 28 additional days are allowed for blood count recovery, if needed.
Period: Overall Study
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Started | 149 | 298
Received Treatment | 149 | 292
Safety Follow Up | 149 (I participant was not treated and 1 participant entered from the Idasanutlin arm) | 292 (5 participants were not treated, 1 participant did not receive Idasanutlin and was moved to the Placebo arm)
Completed | 0 | 0
Not Completed | 149 | 298
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Death | 109 | 211
Not completed — Did not complete due to 2 ineligibilities and physician's decision | 0 | 3
Not completed — Study Terminated By Sponsor | 33 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine | Total
Number analyzed (Participants) | 149 | 298 | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (12.1) | 59.4 (13.1) | 59.6 (12.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 86 | 163 | 249
  Female | 63 | 135 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 112 | 231 | 343
  Not Stated | 18 | 36 | 54
  Unknown | 11 | 20 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 11 | 20 | 31
  Black or African America | 2 | 4 | 6
  Native Hawaiian or other | 0 | 1 | 1
  White | 111 | 222 | 333
  Unknown | 25 | 51 | 76

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in TP53 WT Population
Description: P53 tumor protein Wild Type (TP53 WT) population's Overall Survival was compared in participants with relapsed or refractory (R/R) acute myeloid leukemia (AML) who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo.
  The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: From randomization to death from any cause (up to approximately 4.5 years)
Population: TP53-WT ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Months | 9.13 [7.59 to 10.64] | 8.28 [6.67 to 10.87]
Statistical Analysis 1: Comparison: Placebo Plus Cytarabine vs Idasanutlin Plus Cytarabine; Test type: Superiority; p = 0.5752, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.81 to 1.45]

2. Secondary Outcome: Percentage of Participants in Complete Response (CR) at the End of Induction According to Hematologic Malignancy Response Assessment (HMRA) in TP53 WT Population
Description: Rate of complete response at the end of induction in the TP53 WT population was compared in participants who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo.
  The design followed a hierarchical statistical testing framework.
Time Frame: At the end of induction (up to Day 56)
Population: TP53-WT ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Percentage of Participants | 20.3 | 17.1

3. Secondary Outcome: Event-Free Survival (EFS) According to HMRA in TP53 WT Population
Description: Event Free Survival (EFS) is defined as the time from the date of randomization to whichever occurs first: treatment failure (failure to achieve CR, set as day of final response assessment), relapse from CR, or death from any cause. The study was terminated because of futility, therefore did not reach the planned end of the study.
  The design followed a hierarchical statistical testing framework.
Time Frame: From randomization up to treatment failure, relapse, or death from any cause (up to approximately 4.5 years)
Population: TP53-WT ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Weeks | 6.29 [5.86 to 8.00] | 4.36 [4.14 to 5.00]

4. Secondary Outcome: Percentage of Participants With Overall Remission (CR, CRp, and CRi) at the End of Induction According to HMRA in TP53 WT Population
Description: Rate of overall remission (complete remission, complete remission with incomplete hematologic recovery, complete remission with incomplete platelet count recovery) at the end of induction in the TP53 WT population was compared in participants who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo.
  The design followed a hierarchical statistical testing framework.
Time Frame: At the end of induction (up to Day 56)
Population: TP53-WT ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Percentage of Participants | 38.8 | 22.0

5. Secondary Outcome: Duration of Remission Following CR (DOR) in TP53 WT Population
Description: DOR is defined for patients achieving complete remission and is the time from clinical remission until relapse or death from any cause, whichever occurs first. For patients with none of these events before time of analysis, DOR is censored at the date of the patient's last response assessment.
  The Median upper limits were set to 999 because they were not reached and therefore it was Not Evaluable (NE) and the field is numeric only. The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: From achieving CR until relapse or death from any cause (up to approximately 4.5 years)
Population: TP53-WT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 25 | 59
Months | 18.73 [5.26 to NA] — Insufficient number of participants with events | 16.76 [7.82 to NA] — Insufficient number of participants with events

6. Secondary Outcome: Percentage of Participants Undergoing HSCT Following Complete Response (CR), in TP53 WT Population
Description: Rate of complete response at the end of induction in mutation-defined subgroups (positive for mutation of FLT3, IDH1 and IDH2, respectively) of the TP53 WT population was compared in participants who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo. The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: Baseline up to approximately 4.5 years
Population: TP53-WT ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Percentage of Participants | 10.6 | 11.6

7. Secondary Outcome: Percentage of Participants With Complete Response (CR) in Clinically Actionable Mutation-Defined Subpopulation (FLT3, IDH1 and IDH2) in TP53 WT Population
Description: Rate of complete response at the end of induction in mutation-defined subgroups (positive for mutation of FLT3, IDH1 and IDH2, respectively) of the TP53 WT population was compared in participants who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo.
Time Frame: At the end of induction (up to Day 56)
Population: TP53-WT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Percentage of Participants
  FLT3: number analyzed (Participants) | 59 | 16
  FLT3 | 12.5 | 15.3
  IDH1: number analyzed (Participants) | 23 | 18
  IDH1 | 11.1 | 34.8
  IDH2: number analyzed (Participants) | 44 | 13
  IDH2 | 23.1 | 29.5

8. Secondary Outcome: Overall Survival in Clinically Actionable Mutation-Defined Subpopulation (FLT3, IDH1 and IDH2) in TP53 WT Population
Description: Overall survival in mutation-defined subgroups (positive for mutation of FLT3, IDH1 and IDH2 respectively) of the TP53 WT population was compared in participants who had been randomized to idasanutlin in combination with cytarabine versus those who had been randomized to cytarabine and placebo. The Median upper limits were set to 999 because they were not reached and therefore it was Not Evaluable (NE) and the field is numeric only. The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: From randomization to death from any cause (up to approximately 4.5 years)
Population: TP53-WT ITT Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 123 | 232
Months
  IDH2: number analyzed (Participants) | 44 | 13
  IDH2 | 11.37 [8.02 to NA] — Insufficient number of participants with events | 11.01 [6.87 to NA] — Insufficient number of participants with events
  IDH1: number analyzed (Participants) | 23 | 18
  IDH1 | 9.13 [2.50 to 16.69] | 8.25 [4.27 to 37.29]
  FLT3: number analyzed (Participants) | 59 | 16
  FLT3 | 4.76 [1.97 to 13.04] | 5.55 [4.50 to 8.25]

9. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 (NCI-CTCAE v4.03)
Description: Participants who experienced at least one Adverse Event by severity, According to National Cancer Institute common terminology criteria for Adverse Events, version 4.03 (NCI-CTCAE v4.03) have been reported. The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: Baseline up to approximately 4.5 years
Population: Safety-Evaluable Population
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants | 149 | 232

10. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: Participants with Adverse Events leading to discontinuation of the study have been reported. The study was terminated because of futility, therefore did not reach the planned end of the study.
Time Frame: Baseline up to approximately 4.5 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events Leading to Death up to Day 30
Description: The number of participants with AE resulted by death within 30 days from dosing is reported
Time Frame: Up to Day 30
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants | 9 | 23

12. Secondary Outcome: Number of Participants With Adverse Events Leading to Death up to Day 60
Description: The number of participants with AE resulted by death within 60 days from dosing is reported
Time Frame: Up to Day 60
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants | 24 | 60

13. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Biochemistry Tests at the Greatest Severity, According to NCI-CTCAE v4.03
Description: Laboratory parameters for blood biochemistry will be measured and compared with a standard reference range. Values outside the standard reference range are considered abnormalities. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment or a medical intervention; or is clinically significant in the investigator's judgment.
  For each patient, baseline is the last observation prior to initiation of study drug. For each laboratory test, patients with at least 1 post-baseline assessment are included in the analysis. For each cell, the denominator is the number of patients with baseline NCI-CTCAE Grade 0-2 in the specified direction of abnormality, or Grade 1-4 in the opposite direction of abnormality.
Time Frame: Up to Approximately 4.5 Years
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants
  Albumin Low: number analyzed (Participants) | 149 | 291
  Albumin Low | 8 | 22
  Alkaline Phosphatase High: number analyzed (Participants) | 148 | 291
  Alkaline Phosphatase High | 2 | 9
  SGPT/ALT High: number analyzed (Participants) | 147 | 292
  SGPT/ALT High | 13 | 16
  SGOT/AST High: number analyzed (Participants) | 147 | 290
  SGOT/AST High | 9 | 13
  Calcium Low: number analyzed (Participants) | 147 | 292
  Calcium Low | 8 | 36
  Creatinine High | 4 | 11
  Glucose Low: number analyzed (Participants) | 145 | 285
  Glucose Low | 1 | 0
  Glucose High: number analyzed (Participants) | 144 | 281
  Glucose High | 9 | 25
  Magnesium Low: number analyzed (Participants) | 148 | 287
  Magnesium Low | 0 | 8
  Magnesium High: number analyzed (Participants) | 146 | 287
  Magnesium High | 5 | 10
  Phosphorus Low: number analyzed (Participants) | 142 | 281
  Phosphorus Low | 18 | 72
  Potassium High | 5 | 8
  Sodium Low: number analyzed (Participants) | 148 | 290
  Sodium Low | 6 | 17
  Sodium High | 1 | 7
  Bilirubin High | 9 | 42
  Uric Acid High: number analyzed (Participants) | 141 | 263
  Uric Acid High | 29 | 53
  Potassium Low: number analyzed (Participants) | 149 | 288
  Potassium Low | 21 | 76

14. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Hematology Tests at the Greatest Severity, According to NCI-CTCAE v4.03
Description: Laboratory parameters for hematology will be measured and compared with a standard reference range. Values outside the standard reference range are considered abnormalities. A laboratory test result will be reported as an adverse event if it meets any of the following criteria: is accompanied by clinical symptoms; results in a change in study treatment or a medical intervention; or is clinically significant in the investigator's judgment.
  For each patient, baseline is the last observation prior to initiation of study drug. For each laboratory test, patients with at least 1 post-baseline assessment are included in the analysis. For each cell, the denominator is the number of patients with baseline NCI-CTCAE Grade 0-2 in the specified direction of abnormality, or Grade 1-4 in the opposite direction of abnormality.
Time Frame: Up to Approximately 4.5 Years
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Participants
  Hemoglobin Low: number analyzed (Participants) | 119 | 239
  Hemoglobin Low | 83 | 191
  Hemoglobin High | 1 | 1
  Lymphocytes Abs Low: number analyzed (Participants) | 129 | 242
  Lymphocytes Abs Low | 109 | 229
  Lymphocytes Abs High: number analyzed (Participants) | 148 | 287
  Lymphocytes Abs High | 1 | 1
  Neutrophils, Total, Abs Low: number analyzed (Participants) | 43 | 100
  Neutrophils, Total, Abs Low | 40 | 97
  Platelet Low: number analyzed (Participants) | 60 | 129
  Platelet Low | 59 | 128
  Total Leukocyte Count Low: number analyzed (Participants) | 95 | 186
  Total Leukocyte Count Low | 87 | 184
  Total Leukocyte Count High: number analyzed (Participants) | 148 | 292
  Total Leukocyte Count High | 1 | 1

15. Secondary Outcome: Change From Baseline in Body Temperature Over Time
Description: Vital signs were measured prior to the infusion while the participant was in a seated position. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
  The study was terminated because of futility, therefore did not reach the planned end of study.
Time Frame: Baseline; Cycles 1-3, Days 8, 15, 22, 28 (1 cycle is 28 days); and, if incomplete blood count recovery, Days 29-42 and Days 43-56, Cycles 2 -3 Days 1, 8, 15, 22, 28 and 29-56 (max delay between cycles is 56 days)
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: C, Celsius Degree
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
C, Celsius Degree
  Baseline | 36.49 (0.59) | 36.52 (0.51)
  Cycle 1 Day 8: number analyzed (Participants) | 145 | 284
  Cycle 1 Day 8 | 0.07 (0.82) | 0.32 (0.72)
  Cycle 1 Day 15: number analyzed (Participants) | 136 | 278
  Cycle 1 Day 15 | 0.30 (0.91) | 0.46 (0.92)
  Cycle 1 Day 22: number analyzed (Participants) | 119 | 255
  Cycle 1 Day 22 | 0.22 (0.74) | 0.36 (0.86)
  Cycle 1 Day 28: number analyzed (Participants) | 92 | 201
  Cycle 1 Day 28 | 0.06 (0.65) | 0.23 (0.87)
  Cycle 1 Day 29-42: number analyzed (Participants) | 44 | 139
  Cycle 1 Day 29-42 | 0.08 (0.69) | 0.00 (0.71)
  Cycle 1 Day 43-56: number analyzed (Participants) | 13 | 54
  Cycle 1 Day 43-56 | -0.02 (0.53) | 0.07 (0.80)
  Cycle 2 Day 1: number analyzed (Participants) | 23 | 50
  Cycle 2 Day 1 | 0.11 (0.60) | -0.10 (0.47)
  Cycle 2 Day 8: number analyzed (Participants) | 21 | 44
  Cycle 2 Day 8 | -0.08 (0.51) | 0.07 (0.56)
  Cycle 2 Day 15: number analyzed (Participants) | 23 | 47
  Cycle 2 Day 15 | 0.17 (0.76) | 0.34 (0.83)
  Cycle 2 Day 22: number analyzed (Participants) | 19 | 41
  Cycle 2 Day 22 | 0.04 (0.72) | 0.10 (0.59)
  Cycle 2 Day 28: number analyzed (Participants) | 16 | 33
  Cycle 2 Day 28 | -0.22 (0.65) | 0.04 (0.62)
  Cycle 2 Day 29-56: number analyzed (Participants) | 9 | 26
  Cycle 2 Day 29-56 | -0.06 (0.36) | -0.09 (0.55)
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 16
  Cycle 3 Day 1 | -0.25 (0.54) | -0.19 (0.51)
  Cycle 3 Day 8: number analyzed (Participants) | 13 | 14
  Cycle 3 Day 8 | 0.10 (0.60) | -0.04 (0.59)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 15
  Cycle 3 Day 15 | -0.09 (0.76) | 0.29 (0.65)
  Cycle 3 Day 22: number analyzed (Participants) | 12 | 14
  Cycle 3 Day 22 | -0.07 (0.64) | 0.04 (0.49)
  Cycle 3 Day 28: number analyzed (Participants) | 10 | 11
  Cycle 3 Day 28 | -0.26 (0.63) | -0.15 (0.52)
  Cycle 3 Day 29-56: number analyzed (Participants) | 3 | 10
  Cycle 3 Day 29-56 | 0.27 (0.47) | -0.25 (0.52)

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Millimeters of mercury (mmHg)
  Baseline | 120.6 (17.2) | 122.1 (16.2)
  Cycle 1 Day 8: number analyzed (Participants) | 146 | 285
  Cycle 1 Day 8 | -3.7 (20.0) | -6.9 (18.6)
  Cycle 1 Day 15: number analyzed (Participants) | 138 | 178
  Cycle 1 Day 15 | -2.8 (19.2) | -0.1 (18.7)
  Cycle 1 Day 22: number analyzed (Participants) | 118 | 254
  Cycle 1 Day 22 | 0.7 (20.3) | -1.5 (19.6)
  Cycle 1 Day 28: number analyzed (Participants) | 94 | 201
  Cycle 1 Day 28 | 1.2 (21.7) | -0.5 (17.6)
  Cycle 1 Day 29-42: number analyzed (Participants) | 45 | 141
  Cycle 1 Day 29-42 | 4.4 (17.8) | 3.4 (17.7)
  Cycle 1 Day 43-56: number analyzed (Participants) | 13 | 54
  Cycle 1 Day 43-56 | 9.8 (17.4) | 3.8 (20.9)
  Cycle 2 Day 1: number analyzed (Participants) | 23 | 50
  Cycle 2 Day 1 | 6.9 (15.6) | 0.6 (15.2)
  Cycle 2 Day 8: number analyzed (Participants) | 21 | 44
  Cycle 2 Day 8 | 5.3 (18.6) | -5.1 (16.2)
  Cycle 2 Day 15: number analyzed (Participants) | 23 | 47
  Cycle 2 Day 15 | -1.7 (17.7) | -0.2 (19.6)
  Cycle 2 Day 22: number analyzed (Participants) | 19 | 41
  Cycle 2 Day 22 | 5.5 (19.8) | 2.5 (17.0)
  Cycle 2 Day 28: number analyzed (Participants) | 16 | 33
  Cycle 2 Day 28 | 5.8 (22.2) | 5.0 (17.9)
  Cycle 2 Day 29-56: number analyzed (Participants) | 9 | 26
  Cycle 2 Day 29-56 | -1.0 (18.2) | 6.6 (16.3)
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 16
  Cycle 3 Day 1 | 11.2 (18.9) | 2.3 (18.2)
  Cycle 3 Day 8: number analyzed (Participants) | 13 | 14
  Cycle 3 Day 8 | 6.0 (23.5) | -1.7 (13.4)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 15
  Cycle 3 Day 15 | 3.3 (22.5) | 0.2 (21.7)
  Cycle 3 Day 22: number analyzed (Participants) | 12 | 14
  Cycle 3 Day 22 | 13.9 (22.8) | -1.1 (17.7)
  Cycle 3 Day 28: number analyzed (Participants) | 10 | 11
  Cycle 3 Day 28 | 5.3 (23.0) | 7.1 (18.0)
  Cycle 3 Day 29-56: number analyzed (Participants) | 3 | 10
  Cycle 3 Day 29-56 | 27.7 (28.3) | 5.1 (18.4)

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Millimeters of mercury (mmHg)
  Baseline | 70.2 (9.9) | 71.5 (10.6)
  Cycle 1 Day 8: number analyzed (Participants) | 146 | 285
  Cycle 1 Day 8 | -1.5 (12.6) | -3.1 (12.7)
  Cycle 1 Day 15: number analyzed (Participants) | 138 | 278
  Cycle 1 Day 15 | -1.3 (11.3) | -1.3 (12.3)
  Cycle 1 Day 22: number analyzed (Participants) | 118 | 254
  Cycle 1 Day 22 | -0.5 (11.1) | -1.4 (12.9)
  Cycle 1 Day 28: number analyzed (Participants) | 94 | 201
  Cycle 1 Day 28 | 1.0 (13.2) | -0.7 (12.6)
  Cycle 1 Day 29-42: number analyzed (Participants) | 45 | 141
  Cycle 1 Day 29-42 | 3.8 (10.5) | 0.6 (12.4)
  Cycle 1 Day 43-56: number analyzed (Participants) | 13 | 54
  Cycle 1 Day 43-56 | 1.7 (11.8) | 0.9 (13.5)
  Cycle 2 Day 1: number analyzed (Participants) | 23 | 50
  Cycle 2 Day 1 | 1.1 (13.5) | 0.9 (12.9)
  Cycle 2 Day 8: number analyzed (Participants) | 21 | 44
  Cycle 2 Day 8 | 0.4 (13.5) | -2.2 (13.2)
  Cycle 2 Day 15: number analyzed (Participants) | 23 | 47
  Cycle 2 Day 15 | -0.6 (14.8) | -1.5 (15.4)
  Cycle 2 Day 22: number analyzed (Participants) | 19 | 41
  Cycle 2 Day 22 | 3.1 (11.6) | 1.7 (11.3)
  Cycle 2 Day 28: number analyzed (Participants) | 16 | 33
  Cycle 2 Day 28 | 4.6 (13.9) | 3.9 (12.7)
  Cycle 2 Day 29-56: number analyzed (Participants) | 9 | 26
  Cycle 2 Day 29-56 | -2.9 (12.4) | 3.2 (15.8)
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 16
  Cycle 3 Day 1 | 5.0 (8.4) | 0.3 (10.7)
  Cycle 3 Day 8: number analyzed (Participants) | 13 | 14
  Cycle 3 Day 8 | 2.0 (15.5) | -3.3 (11.8)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 15
  Cycle 3 Day 15 | 0.7 (11.1) | -1.8 (11.1)
  Cycle 3 Day 22: number analyzed (Participants) | 12 | 14
  Cycle 3 Day 22 | 10.1 (14.3) | -2.1 (9.3)
  Cycle 3 Day 28: number analyzed (Participants) | 10 | 11
  Cycle 3 Day 28 | 2.3 (14.7) | 1.3 (10.1)
  Cycle 3 Day 29-56: number analyzed (Participants) | 3 | 10
  Cycle 3 Day 29-56 | 5.0 (21.8) | 2.6 (13.6)

18. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Beats per Minute
  Baseline | 78.4 (14.4) | 79.2 (12.9)
  Cycle 1 Day 8: number analyzed (Participants) | 145 | 283
  Cycle 1 Day 8 | -4.3 (15.9) | 3.4 (15.6)
  Cycle 1 Day 15: number analyzed (Participants) | 138 | 278
  Cycle 1 Day 15 | 1.5 (16.0) | 1.1 (17.2)
  Cycle 1 Day 22: number analyzed (Participants) | 116 | 253
  Cycle 1 Day 22 | 0.2 (16.2) | 4.1 (15.8)
  Cycle 1 Day 28: number analyzed (Participants) | 94 | 197
  Cycle 1 Day 28 | 4.8 (15.8) | 4.0 (16.8)
  Cycle 1 Day 29-42: number analyzed (Participants) | 25 | 141
  Cycle 1 Day 29-42 | 2.0 (13.5) | 5.1 (16.4)
  Cycle 1 Day 43-56: number analyzed (Participants) | 13 | 53
  Cycle 1 Day 43-56 | 5.5 (18.6) | 6.8 (14.0)
  Cycle 2 Day 1: number analyzed (Participants) | 23 | 50
  Cycle 2 Day 1 | 2.0 (16.6) | -0.9 (12.0)
  Cycle 2 Day 8: number analyzed (Participants) | 21 | 42
  Cycle 2 Day 8 | -3.3 (18.6) | 2.4 (14.9)
  Cycle 2 Day 15: number analyzed (Participants) | 23 | 47
  Cycle 2 Day 15 | -0.4 (12.7) | 1.7 (18.4)
  Cycle 2 Day 22: number analyzed (Participants) | 19 | 40
  Cycle 2 Day 22 | 2.3 (15.5) | 0.3 (15.4)
  Cycle 2 Day 28: number analyzed (Participants) | 16 | 31
  Cycle 2 Day 28 | -2.3 (14.6) | 1.2 (12.2)
  Cycle 2 Day 29-56: number analyzed (Participants) | 9 | 26
  Cycle 2 Day 29-56 | 1.8 (11.8) | 4.0 (14.8)
  Cycle 3 Day 1: number analyzed (Participants) | 15 | 16
  Cycle 3 Day 1 | 0.4 (18.4) | 1.0 (9.8)
  Cycle 3 Day 8: number analyzed (Participants) | 13 | 13
  Cycle 3 Day 8 | 1.3 (21.5) | 2.4 (16.2)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 15
  Cycle 3 Day 15 | 2.5 (16.9) | 1.9 (11.9)
  Cycle 3 Day 22: number analyzed (Participants) | 12 | 14
  Cycle 3 Day 22 | 4.8 (19.7) | 3.4 (13.6)
  Cycle 3 Day 28: number analyzed (Participants) | 10 | 11
  Cycle 3 Day 28 | 0.4 (16.1) | 0.9 (13.7)
  Cycle 3 Day 29-56: number analyzed (Participants) | 3 | 10
  Cycle 3 Day 29-56 | -5.0 (1.7) | 5.2 (11.5)

19. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Description: as for outcome 15
Time Frame: Up to Approximately 4.5 Years
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Breaths per Minute
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Breaths per Minute
  Baseline: number analyzed (Participants) | 134 | 261
  Baseline | 16.3 (2.7) | 16.6 (2.7)
  Cycle 1 Day 8: number analyzed (Participants) | 101 | 200
  Cycle 1 Day 8 | -0.1 (2.7) | 0.0 (2.8)
  Cycle 1 Day 15: number analyzed (Participants) | 94 | 186
  Cycle 1 Day 15 | 0.7 (2.9) | 0.4 (2.8)
  Cycle 1 Day 22: number analyzed (Participants) | 77 | 169
  Cycle 1 Day 22 | 0.6 (3.2) | 0.7 (4.1)
  Cycle 1 Day 28: number analyzed (Participants) | 70 | 130
  Cycle 1 Day 28 | 0.4 (2.9) | 0.6 (2.9)
  Cycle 1 Day 29-42: number analyzed (Participants) | 33 | 96
  Cycle 1 Day 29-42 | 0.7 (2.1) | 0.5 (2.7)
  Cycle 1 Day 43-56: number analyzed (Participants) | 9 | 38
  Cycle 1 Day 43-56 | 0.3 (1.0) | 0.0 (2.9)
  Cycle 2 Day 1: number analyzed (Participants) | 17 | 35
  Cycle 2 Day 1 | -0.3 (2.8) | -0.2 (3.2)
  Cycle 2 Day 8: number analyzed (Participants) | 13 | 28
  Cycle 2 Day 8 | -0.2 (2.9) | 0.1 (3.3)
  Cycle 2 Day 15: number analyzed (Participants) | 15 | 28
  Cycle 2 Day 15 | 0.5 (2.4) | 0.0 (2.5)
  Cycle 2 Day 22: number analyzed (Participants) | 13 | 23
  Cycle 2 Day 22 | 0.8 (2.3) | 0.4 (1.4)
  Cycle 2 Day 28: number analyzed (Participants) | 12 | 23
  Cycle 2 Day 28 | -0.3 (2.3) | 0.5 (3.5)
  Cycle 2 Day 29-56: number analyzed (Participants) | 5 | 22
  Cycle 2 Day 29-56 | 0.2 (1.8) | 0.3 (2.5)
  Cycle 3 Day 1: number analyzed (Participants) | 11 | 11
  Cycle 3 Day 1 | 1.1 (2.5) | 0.2 (2.1)
  Cycle 3 Day 8: number analyzed (Participants) | 10 | 11
  Cycle 3 Day 8 | 0.2 (2.5) | -1.0 (3.1)
  Cycle 3 Day 15: number analyzed (Participants) | 11 | 9
  Cycle 3 Day 15 | 1.5 (3.6) | 0.9 (2.2)
  Cycle 3 Day 22: number analyzed (Participants) | 8 | 9
  Cycle 3 Day 22 | 1.1 (2.7) | 0.8 (1.6)
  Cycle 3 Day 28: number analyzed (Participants) | 8 | 8
  Cycle 3 Day 28 | 0.3 (1.2) | 0.8 (1.8)
  Cycle 3 Day 29-56: number analyzed (Participants) | 3 | 7
  Cycle 3 Day 29-56 | 0.7 (4.6) | 0.1 (2.4)

20. Secondary Outcome: Change From Baseline in Heart Rate, as Measured by Electrocardiogram
Description: Single 12-lead ECGs was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. The baseline value at visit and the change from baseline value at each timepoint are reported. The change from baseline value was calculated by subtracting the post-baseline value from the baseline value.
  The study was terminated because of futility, therefore did not reach the planned end of study.
Time Frame: Baseline; Cycles 1-3 Day 1 (2 hrs pre-dose, post-Cytarabine and 6 hrs post-Idasanutlin/Placebo ); Cycle 1-3 Day 2; Cycle 1 Day 5 (within 2 hrs Idanasanutlin/Placebo, post-Cytarabine and 6 hrs post-Idasanutlin/Placebo), Study Drug Completion
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Beats per Minute
  Baseline: number analyzed (Participants) | 149 | 286
  Baseline | 77.3 (13.2) | 78.6 (14.2)
  Cycle 1 Day 1 2 Hours Pre-dose: number analyzed (Participants) | 16 | 40
  Cycle 1 Day 1 2 Hours Pre-dose | 1.1 (11.6) | -0.8 (11.7)
  Cycle 1 Day 1 Post-Cytarabine: number analyzed (Participants) | 144 | 273
  Cycle 1 Day 1 Post-Cytarabine | -0.1 (8.4) | -0.4 (9.8)
  Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 142 | 269
  Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | 0.1 (9.6) | 1.4 (9.2)
  Cycle 1 Day 2: number analyzed (Participants) | 143 | 274
  Cycle 1 Day 2 | -2.2 (11.0) | -0.4 (11.7)
  Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 142 | 271
  Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | -10.3 (14.4) | -1.2 (14.3)
  Cycle 1 Day 5 - Post-Cytarabine: number analyzed (Participants) | 133 | 263
  Cycle 1 Day 5 - Post-Cytarabine | -9.9 (12.8) | -3.0 (14.2)
  Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 135 | 232
  Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | -10.7 (13.2) | -3.1 (14.0)
  Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 10 | 28
  Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -0.5 (13.5) | -4.8 (12.0)
  Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 8 | 26
  Cycle 2 Day 1 Post-Cytarabine | 0.8 (17.3) | -4.8 (12.6)
  Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 21
  Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | -0.7 (16.6) | -0.7 (15.6)
  Cycle 2 Day 2: number analyzed (Participants) | 8 | 23
  Cycle 2 Day 2 | -5.2 (15.7) | -4.8 (10.3)
  Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 6
  Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -3.0 (14.2) | -7.1 (10.2)
  Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  Cycle 3 Day 1 Post-Cytarabine | -8.9 (21.0) | -4.5 (7.4)
  Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | -2.0 (17.2) | -0.1 (15.0)
  Cycle 3 Day 2: number analyzed (Participants) | 5 | 5
  Cycle 3 Day 2 | 0.1 (14.7) | -9.3 (8.8)
  Study Drug Completion/Discontinuation: number analyzed (Participants) | 81 | 145
  Study Drug Completion/Discontinuation | 3.4 (15.9) | 4.5 (16.4)

21. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters: PQ, PR, RR, QRS, QT and QTcF Intervals
Description: as for outcome 20
Time Frame: Baseline, Days 1, 2, and 5 of Cycle 1, Days 1, 2 of Cycles 2 and 3 (1 cycle is 28 days), Treatment Discontinuation Visit (28 days after last dose of study drug)
Population: Safety Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Millisecond (msec)
  PR Duration Baseline: number analyzed (Participants) | 148 | 281
  PR Duration Baseline | 160.3 (37.5) | 155.5 (32.4)
  PR Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 16 | 41
  PR Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 12.4 (54.8) | -2.7 (52.6)
  PR Duration Cycle 1 Day 1 - Post-Cytarabine: number analyzed (Participants) | 142 | 269
  PR Duration Cycle 1 Day 1 - Post-Cytarabine | 4.8 (40.9) | 1.6 (30.4)
  PR Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 139 | 265
  PR Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | 0.6 (46.0) | 1.6 (28.4)
  PR Duration Cycle 1 Day 2: number analyzed (Participants) | 141 | 268
  PR Duration Cycle 1 Day 2 | 2.1 (28.8) | 1.4 (25.8)
  PR Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 138 | 261
  PR Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | -3.0 (31.5) | -2.1 (25.0)
  PR Duration Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 130 | 256
  PR Duration Cycle 1 Day 5 Post-Cytarabine | 1.2 (50.3) | -1.6 (18.3)
  PR Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 133 | 253
  PR Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | -5.7 (30.3) | -3.5 (24.6)
  PR Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 10 | 28
  PR Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 30.0 (75.9) | 2.2 (17.6)
  PR Duration Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 8 | 26
  PR Duration Cycle 2 Day 1 Post-Cytarabine | -4.2 (15.2) | 4.9 (11.7)
  PR Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 21
  PR Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | -3.0 (16.8) | 6.0 (14.6)
  PR Duration Cycle 2 Day 2: number analyzed (Participants) | 8 | 23
  PR Duration Cycle 2 Day 2 | -3.0 (18.7) | 5.9 (12.3)
  PR Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 6
  PR Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 9.3 (28.6) | 6.7 (11.7)
  PR Duration Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  PR Duration Cycle 3 Day 1 Post-Cytarabine | -7.7 (5.3) | 3.9 (10.0)
  PR Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  PR Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | -4.5 (9.9) | 6.9 (12.0)
  PR Duration Cycle 3 Day 2: number analyzed (Participants) | 5 | 5
  PR Duration Cycle 3 Day 2 | -1.0 (3.3) | 14.1 (12.9)
  PR Duration Study Drug Completion/Discontinuation: number analyzed (Participants) | 79 | 140
  PR Duration Study Drug Completion/Discontinuation | -5.3 (28.6) | -7.7 (37.1)
  QRS Duration Baseline: number analyzed (Participants) | 149 | 286
  QRS Duration Baseline | 92.8 (17.7) | 89.3 (16.5)
  QRS Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 16 | 41
  QRS Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -0.4 (3.2) | -1.9 (6.2)
  QRS Duration Cycle 1 Day 1 Post-Cytarabine: number analyzed (Participants) | 142 | 274
  QRS Duration Cycle 1 Day 1 Post-Cytarabine | -0.9 (10.0) | -1.0 (6.7)
  QRS Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 141 | 270
  QRS Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | -0.6 (18.4) | -1.1 (6.9)
  QRS Duration Cycle 1 Day 2: number analyzed (Participants) | 142 | 273
  QRS Duration Cycle 1 Day 2 | -0.5 (11.6) | 1.1 (7.8)
  QRS Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 140 | 268
  QRS Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | 1.1 (8.7) | 1.6 (9.1)
  QRS Duration Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 131 | 261
  QRS Duration Cycle 1 Day 5 Post-Cytarabine | 0.6 (12.2) | 0.2 (11.2)
  QRS Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 134 | 261
  QRS Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | 0.3 (13.0) | -0.3 (10.6)
  QRS Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 10 | 28
  QRS Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 0.8 (4.7) | 0.4 (8.0)
  QRS Duration Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 8 | 26
  QRS Duration Cycle 2 Day 1 Post-Cytarabine | 6.5 (12.2) | -2.1 (9.4)
  QRS Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 21
  QRS Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | 2.0 (13.9) | 0.1 (6.6)
  QRS Duration Cycle 2 Day 2: number analyzed (Participants) | 7 | 23
  QRS Duration Cycle 2 Day 2 | 0.3 (6.3) | 0.2 (7.1)
  QRS Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 6
  QRS Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -0.1 (5.9) | -2.4 (5.9)
  QRS Duration Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  QRS Duration Cycle 3 Day 1 Post-Cytarabine | 2.7 (5.3) | -2.0 (3.4)
  QRS Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  QRS Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | 0.4 (5.4) | -2.7 (3.8)
  QRS Duration Cycle 3 Day 2: number analyzed (Participants) | 5 | 5
  QRS Duration Cycle 3 Day 2 | 1.5 (6.6) | -1.6 (8.7)
  QRS Duration Study Drug Completion/Discontinuation: number analyzed (Participants) | 81 | 146
  QRS Duration Study Drug Completion/Discontinuation | -1.3 (10.1) | -0.4 (12.7)
  QT Duration Baseline: number analyzed (Participants) | 149 | 286
  QT Duration Baseline | 388.7 (35.9) | 385.6 (35.7)
  QT Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 16 | 41
  QT Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 6.0 (30.6) | 4.2 (32.4)
  QT Duration Cycle 1 Day 1 Post-Cytarabine: number analyzed (Participants) | 143 | 274
  QT Duration Cycle 1 Day 1 Post-Cytarabine | 0.7 (25.3) | 4.4 (24.2)
  QT Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 140 | 270
  QT Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | 1.1 (28.2) | 0.0 (25.4)
  QT Duration Cycle 1 Day 2: number analyzed (Participants) | 142 | 247
  QT Duration Cycle 1 Day 2 | 5.4 (31.9) | 3.1 (31.7)
  QT Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 140 | 269
  QT Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | 24.8 (44.6) | 1.6 (35.5)
  QT Duration Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 132 | 232
  QT Duration Cycle 1 Day 5 Post-Cytarabine | 25.0 (41.0) | 4.7 (36.6)
  QT Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 134 | 232
  QT Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | 27.8 (42.3) | 3.4 (34.8)
  QT Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 10 | 28
  QT Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -9.1 (34.8) | 8.5 (31.3)
  QT Duration Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 8 | 26
  QT Duration Cycle 2 Day 1 Post-Cytarabine | -11.5 (29.2) | 10.6 (31.3)
  QT Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 21
  QT Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | -7.5 (31.4) | 4.1 (39.7)
  QT Duration Cycle 2 Day 2: number analyzed (Participants) | 7 | 23
  QT Duration Cycle 2 Day 2 | 12.2 (24.7) | 9.9 (38.6)
  QT Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 6
  QT Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 1.9 (33.4) | 15.9 (33.8)
  QT Duration Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  QT Duration Cycle 3 Day 1 Post-Cytarabine | 21.2 (33.2) | 22.0 (35.3)
  QT Duration Cycle 3 Day 1 - 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  QT Duration Cycle 3 Day 1 - 6 Hours Post-Idasanutlin/Placebo | -3.4 (32.2) | 19.0 (34.2)
  QT Duration Cycle 3 Day 2: number analyzed (Participants) | 5 | 5
  QT Duration Cycle 3 Day 2 | -9.4 (13.6) | 28.0 (35.3)
  QT Duration Study Drug Completion/Discontinuation: number analyzed (Participants) | 81 | 146
  QT Duration Study Drug Completion/Discontinuation | -5.6 (36.2) | -4.8 (34.8)
  QTcB Baseline: number analyzed (Participants) | 127 | 243
  QTcB Baseline | 435.3 (30.9) | 437.5 (31.1)
  QTcB Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 14 | 32
  QTcB Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 8.7 (20.5) | 4.8 (23.9)
  QTcB Cycle 1 Day 1 Post-Cytarabin: number analyzed (Participants) | 119 | 223
  QTcB Cycle 1 Day 1 Post-Cytarabin | 1.3 (192) | 3.8 (26.1)
  QTcB Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 117 | 221
  QTcB Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | 1.4 (24.8) | 6.4 (39.5)
  QTcB Cycle 1 Day 2: number analyzed (Participants) | 117 | 220
  QTcB Cycle 1 Day 2 | -1.8 (22.8) | 2.4 (25.9)
  QTcB Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placeb: number analyzed (Participants) | 118 | 217
  QTcB Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placeb | -8.3 (26.2) | -3.2 (27.9)
  QTcB Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 109 | 211
  QTcB Cycle 1 Day 5 Post-Cytarabine | -4.4 (28.7) | -3.7 (23.4)
  QTcB Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 109 | 214
  QTcB Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | -5.2 (28.8) | -5.5 (24.0)
  QTcB Cycle 2 Day 1 - Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 22
  QTcB Cycle 2 Day 1 - Within 2 Hours Pre-Idasanutlin/Placebo | 0.5 (15.7) | 1.6 (32.0)
  QTcB Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 6 | 20
  QTcB Cycle 2 Day 1 Post-Cytarabine | 3.0 (24.8) | 4.2 (45.0)
  QTcB Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 7 | 16
  QTcB Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | 6.5 (27.7) | 4.6 (28.3)
  QTcB Cycle 2 Day 2: number analyzed (Participants) | 6 | 18
  QTcB Cycle 2 Day 2 | 0.8 (28.6) | -1.0 (25.6)
  QTcB Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 6
  QTcB Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 13.1 (24.3) | -1.1 (17.8)
  QTcB Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  QTcB Cycle 3 Day 1 Post-Cytarabine | 16.6 (27.3) | 13.6 (21.4)
  QTcB Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  QTcB Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | 6.9 (24.6) | 21.9 (28.6)
  QTcB Cycle 3 Day 2: number analyzed (Participants) | 5 | 4
  QTcB Cycle 3 Day 2 | 1.4 (18.5) | 14.3 (18.4)
  QTcB Study Drug Completion/Discontinuation: number analyzed (Participants) | 64 | 114
  QTcB Study Drug Completion/Discontinuation | 1.9 (32.2) | 5.8 (29.9)
  QTcF Baseline: number analyzed (Participants) | 127 | 243
  QTcF Baseline | 418.0 (28.5) | 419.0 (26.6)
  QTcF Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 14 | 32
  QTcF Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 7.6 (19.3) | 5.1 (21.7)
  QTcF Cycle 1 Day 1 Post-Cytarabine: number analyzed (Participants) | 119 | 223
  QTcF Cycle 1 Day 1 Post-Cytarabine | 1.0 (18.3) | 4.1 (22.0)
  QTcF Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 117 | 221
  QTcF Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | 0.9 (23.4) | 4.2 (28.6)
  QTcF Cycle 1 Day 2: number analyzed (Participants) | 117 | 220
  QTcF Cycle 1 Day 2 | 1.3 (22.7) | 2.6 (23.8)
  QTcF Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 118 | 217
  QTcF Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | 3.6 (23.7) | -1.1 (24.3)
  QTcF Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 109 | 211
  QTcF Cycle 1 Day 5 Post-Cytarabine | 6.1 (27.1) | -0.4 (22.6)
  QTcF Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 109 | 214
  QTcF Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | 6.0 (27.7) | -2.1 (22.2)
  QTcF Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 22
  QTcF Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 0.0 (19.7) | 4.0 (26.3)
  QTcF Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 6 | 20
  QTcF Cycle 2 Day 1 Post-Cytarabine | 0.5 (15.7) | 6.4 (36.9)
  QTcF Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 7 | 16
  QTcF Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | 1.5 (21.1) | 4.0 (26.8)
  QTcF Cycle 2 Day 2: number analyzed (Participants) | 6 | 18
  QTcF Cycle 2 Day 2 | 6.1 (18.3) | 1.1 (26.3)
  QTcF Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 6
  QTcF Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 14.0 (21.6) | 14.0 (21.6)
  QTcF Cycle 3 Day 1 - Post-Cytarabine: number analyzed (Participants) | 4 | 5
  QTcF Cycle 3 Day 1 - Post-Cytarabine | 18.5 (24.1) | 16.8 (26.0)
  QTcF Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  QTcF Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | 3.5 (25.2) | 20.7 (24.7)
  QTcF Cycle 3 Day 2: number analyzed (Participants) | 5 | 4
  QTcF Cycle 3 Day 2 | -2.6 (14.5) | 19.2 (25.6)
  QTcF Study Drug Completion/Discontinuation: number analyzed (Participants) | 64 | 114
  QTcF Study Drug Completion/Discontinuation | 0.2 (28.3) | 2.9 (26.5)
  RR Duration Baseline: number analyzed (Participants) | 127 | 243
  RR Duration Baseline | 797.9 (139.6) | 787.9 (151.7)
  RR Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 14 | 32
  RR Duration Cycle 1 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -2.5 (63.5) | 4.8 (139.1)
  RR Duration Cycle 1 Day 1 Post-Cytarabine: number analyzed (Participants) | 119 | 223
  RR Duration Cycle 1 Day 1 Post-Cytarabine | -4.7 (89.6) | 3.6 (105.6)
  RR Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 117 | 221
  RR Duration Cycle 1 Day 1 6 Hours Post-Idasanutlin/Placebo | -3.0 (103.4) | -19.1 (108.5)
  RR Duration Cycle 1 Day 2: number analyzed (Participants) | 117 | 220
  RR Duration Cycle 1 Day 2 | 37.6 (117.6) | 4.1 (126.7)
  RR Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 118 | 117
  RR Duration Cycle 1 Day 5 Within 2 Hours Pre-Idasanutlin/Placebo | 159.3 (212.4) | 19.5 (146.8)
  RR Duration Cycle 1 Day 5 Post-Cytarabine: number analyzed (Participants) | 109 | 211
  RR Duration Cycle 1 Day 5 Post-Cytarabine | 133.7 (164.9) | 36.8 (151.5)
  RR Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 109 | 214
  RR Duration Cycle 1 Day 5 6 Hours Post-Idasanutlin/Placebo | 144.2 (167.6) | 37.8 (150.5)
  RR Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 8 | 22
  RR Duration Cycle 2 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | -5.4 (119.6) | 25.7 (156.7)
  RR Duration Cycle 2 Day 1 Post-Cytarabine: number analyzed (Participants) | 6 | 20
  RR Duration Cycle 2 Day 1 Post-Cytarabine | -38.8 (140.1) | 23.3 (123.3)
  RR Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 7 | 16
  RR Duration Cycle 2 Day 1 6 Hours Post-Idasanutlin/Placebo | -66.9 (176.4) | -15.2 (180.8)
  RR Duration Cycle 2 Day 2: number analyzed (Participants) | 6 | 18
  RR Duration Cycle 2 Day 2 | 57.9 (162.2) | 14.1 (155.4)
  RR Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 6
  RR Duration Cycle 3 Day 1 Within 2 Hours Pre-Idasanutlin/Placebo | 15.1 (80.8) | 65.5 (105.1)
  RR Duration Cycle 3 Day 1 Post-Cytarabine: number analyzed (Participants) | 4 | 5
  RR Duration Cycle 3 Day 1 Post-Cytarabine | 11.1 (132.8) | 38.9 (75.0)
  RR Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo: number analyzed (Participants) | 6 | 5
  RR Duration Cycle 3 Day 1 6 Hours Post-Idasanutlin/Placebo | -49.4 (89.8) | 3.3 (135.5)
  RR Duration Cycle 3 Day 2: number analyzed (Participants) | 5 | 4
  RR Duration Cycle 3 Day 2 | -42.9 (72.0) | 62.0 (120.3)
  RR Duration Study Drug Completion/Discontinuation: number analyzed (Participants) | 64 | 114
  RR Duration Study Drug Completion/Discontinuation | -14.8 (170.6) | -14.8 (170.6)

22. Secondary Outcome: Total Duration of Study Treatment
Description: Participants were planned to be treated up to 3 Cycles.
Time Frame: Up to 3 cycles (1 cycle is 28 days)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Idasanutlin Plus Cytarabine | Placebo Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Days | 16.5 (28.29) | 17.6 (28.25)

23. Secondary Outcome: Number of Treatment Cycles Started
Description: Participants who started the study treatment cycles are reported.
Time Frame: Up to 3 cycles (1 cycle is 28 days)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Treatment Cycles
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Treatment Cycles | 1.3 (0.63) | 1.2 (0.54)

24. Secondary Outcome: Cumulative Dose of Idasanutlin and Cytarabine
Description: The cumulative doses of idasanutlin and cytaradine are reported.
Time Frame: Up to 3 cycles (1 cycle is 28 days)
Population: Safety Population. Participants did not receive Idasanutlin in the "Placebo Plus Cytarabine" Arm, so this data were not collected.
Measure: Mean (Standard Deviation); unit: Milligram (mg)
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 149 | 292
Milligram (mg)
  Idasanutlin/Placebo cumulative dose (mg): number analyzed (Participants) | 0 | 292
  Idasanutlin/Placebo cumulative dose (mg) |  | 3340.1 (896.35)
  Cytarabine cumulative dose (mg) | 11500 (5850) | 11200 (5190)

25. Secondary Outcome: Apparent Clearance (CL/F) of Idasanutlin
Description: Apparent Clearance (CL/F) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population. The planned CL/F did not derive for the result data and was not reported.
Time Frame: Cycle 1: Predose (0 hour [Hr]), end of 1-3 Hr cytarabine infusion, 6 Hr postdose on Days 1, 5; Predose (0 Hr) on Day 2; at Days 8, 10; Cycle 2, 3: predose (0 Hr) on Days 2, 5 (predose/postdose: relative to idasanutlin morning dose; cycle length= 28 days)
Population: Due to futility the planned participant enrollment was observed, therefore result data were not collected.
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Idasanutlin
Description: Apparent Volume of Distribution (Vd/F) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: Cycle 1: Predose (0 Hr), end of 1-3 Hr cytarabine infusion, 6 Hr postdose on Days 1, 5; Predose (0 Hr) on Day 2; at Days 8, 10; Cycle 2, 3: predose (0 Hr) on Days 2, 5 (predose/postdose: relative to idasanutlin morning dose; cycle length= 28 days)
Population: Due to insufficient participant compliance the planned enrollment was observed, therefore result data were not collected.
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Maximum Concentration Observed (Cmax) of Idasanutlin
Description: Maximum Concentration Observed (Cmax) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 26
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Steady-State Concentration (Ctrough) of Idasanutlin
Description: Steady-State Concentration (Ctrough) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 26
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) During One Dosing Interval (AUCtau) of Idasanutlin
Description: Area Under the Concentration-Time Curve (AUC) During One Dosing Interval (AUCtau) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 26
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: AUC From Time Zero to 24 Hours Post Dose (AUC0-24) of Idasanutlin
Description: AUC from Time Zero to 24 Hours Post Dose (AUC0-24) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 26
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Half-Life (t 1/2) of Idasanutlin
Description: Half-Life (t 1/2) of Idasanutlin was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 26
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Total Clearance (CL) of Cytarabine
Description: The Total Clearance (CL) of Cytarabine was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: Cycle 1: Within 2 Hr pre-cytarabine dose, end of 1-3 Hr cytarabine infusion, 6 Hr post idasanutlin morning dose on Days 1, 5; Within 2 Hr pre-cytarabine dose on Day 2; Cycle 2, 3: Within 2 Hr pre-cytarabine dose on Day 2 (Cycle length= 28 days)
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Volume of Distribution (Vd) of Cytarabine
Description: The Volume of Distribution (Vd) of Cytarabine was planned as part of the PK analyses. The Independent Data Monitoring Committee recommended stopping the study for futility based on a lack of OS benefit due to Hazard Ratio (HR) being greater than 1. The benefit-risk profile of idasanutlin combined with 1g/m2 cytarabine in fit R/R AML was not positive, as the observed marginal benefit does not outweigh the risks of idasanutlin in the relapsed or refractory AML population.
  Therefore the study was prematurely terminated by the sponsor's decision and the result data did not derive.
Time Frame: as for outcome 32
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Change From Baseline in European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score
Description: The compliance rate (defined as the number of patients who completed as least 1 question on the measure) at baseline was 56% and 61% for the Idasanutlin arm and the placebo arm, respectively. This compliance rate remained the same post-baseline in both arms. Due to the low compliance rates in both arms during the entire treatment period, the planned analyses were not performed.
Time Frame: Cycle 1 Day 1 (Baseline), Days 8, 15, 28 of Cycle 1, Days 1, 8, 15, 28 of Cycles 2, 3, 28 days after last dose (last dose on Cycle 3 Day 5), thereafter every 3 months until relapse (maximum up to 3.5 years)
Population: Due to insufficient participant compliance rate, an insufficient enrollment was observed and result data were not collected.
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5-Level (EQ-5D-5L) Questionnaire Score
Description: The compliance rate (defined as the number of patients who completed as least 1 question on the measure) at baseline was 56% and 61% for the Idasanutlin arm and the placebo arm, respectively. Compliance remained the same post-baseline in both arms Due to the low compliance rates in both arms during the entire treatment period, the planned analyses were not performed.
Time Frame: as for outcome 34
Population: as for outcome 26
Arm/Group | Placebo Plus Cytarabine | Idasanutlin Plus Cytarabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The timeframe was planned to be from the Baseline up to approximately 4.5 years. The study was pre-maturely terminated due to mild benefit by the sponsor's decision, therefore did not reach the planned end of study.
Description: Reported: Safety Evaluable Population. During the Safety Follow-up Period, non-Serious Adverse Events occurred at the 5% frequency threshold.
  In Idasanutlin-Cytarabine Arm, total of 298 participants were enrolled of but 5 participants were not treated, 1 participant did not receive Idasanutlin and was moved to the Placebo Arm. In Placebo Arm, total 149 participants were enrolled,1 participant was not treated and 1 participant entered from the Idasanutlin Arm.
Groups:
- Idasanutlin-Cytarabine: Participants will receive induction therapy idasanutlin and cytarabine for 5 days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or complete remission with incomplete blood count recovery (CRi), up to 28 additional days are allowed for blood count recovery, if needed
- Placebo-Cytarabine: Participants will receive induction therapy idasanutlin matching placebo and cytarabine for 5 days followed by 23 days of rest in Cycle 1 (treatment cycle length=28 days). Responding participants may continue with consolidation therapy for a maximum of 2 additional cycles including idasanutlin matching placebo and cytarabine for 5 days followed by 23 days of rest in each cycle (treatment cycle length=28 days). After each cycle, for participants achieving CRp or CRi, up to 28 additional days are allowed for blood count recovery, if needed.
Arm/Group | Idasanutlin-Cytarabine | Placebo-Cytarabine
All-Cause Mortality (participants affected / at risk) | 211/292 | 109/149
Serious Adverse Events (participants affected / at risk) | 173/292 | 72/149
Other Adverse Events (participants affected / at risk) | 290/292 | 147/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idasanutlin-Cytarabine (N=292) | Placebo-Cytarabine (N=149)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (37) | 13 (16)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 6 (7) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 (6) | 1 (1)
Ocular icterus (Hepatobiliary disorders) | 1 (1) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Chronic graft versus host disease (Immune system disorders) | 1 (1) | 1 (1)
Graft versus host disease (Immune system disorders) | 4 (4) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 3 (3) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 2 (3) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 4 (5) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 2 (2) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Fusobacterium infection (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 5 (6) | 2 (2)
Periorbital cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 21 (21) | 13 (13)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 34 (34) | 8 (8)
Septic shock (Infections and infestations) | 11 (11) | 8 (8)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atypical mycobacterium test positive (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 5 (7) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idasanutlin-Cytarabine (N=292) | Placebo-Cytarabine (N=149)
Anaemia (Blood and lymphatic system disorders) | 79 (131) | 49 (71)
Febrile neutropenia (Blood and lymphatic system disorders) | 136 (178) | 63 (79)
Neutropenia (Blood and lymphatic system disorders) | 35 (36) | 13 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 120 (175) | 69 (104)
Atrial fibrillation (Cardiac disorders) | 15 (20) | 6 (8)
Tachycardia (Cardiac disorders) | 16 (17) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 54 (68) | 18 (19)
Abdominal pain upper (Gastrointestinal disorders) | 24 (28) | 6 (6)
Constipation (Gastrointestinal disorders) | 53 (76) | 76 (99)
Diarrhoea (Gastrointestinal disorders) | 251 (404) | 49 (65)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 15 (19) | 10 (12)
Haemorrhoids (Gastrointestinal disorders) | 18 (22) | 8 (8)
Nausea (Gastrointestinal disorders) | 153 (227) | 47 (56)
Stomatitis (Gastrointestinal disorders) | 24 (24) | 6 (8)
Vomiting (Gastrointestinal disorders) | 89 (145) | 27 (30)
Asthenia (General disorders) | 56 (70) | 19 (24)
Chest pain (General disorders) | 19 (25) | 9 (9)
Fatigue (General disorders) | 28 (30) | 13 (15)
Mucosal inflammation (General disorders) | 46 (50) | 10 (11)
Oedema (General disorders) | 22 (24) | 5 (6)
Oedema peripheral (General disorders) | 65 (88) | 26 (34)
Pyrexia (General disorders) | 108 (174) | 49 (67)
Hyperbilirubinaemia (Hepatobiliary disorders) | 52 (56) | 12 (15)
Bacteraemia (Infections and infestations) | 15 (15) | 2 (2)
Device related infection (Infections and infestations) | 16 (16) | 8 (8)
Oral herpes (Infections and infestations) | 22 (23) | 11 (11)
Pneumonia (Infections and infestations) | 18 (18) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 14 (21) | 10 (11)
Alanine aminotransferase increased (Investigations) | 15 (20) | 12 (12)
Blood creatinine increased (Investigations) | 10 (12) | 9 (10)
Gamma-glutamyltransferase increased (Investigations) | 15 (16) | 9 (9)
Weight increased (Investigations) | 16 (16) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 54 (58) | 14 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 17 (23) | 9 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (23) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 35 (42) | 7 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 129 (207) | 48 (65)
Hypomagnesaemia (Metabolism and nutrition disorders) | 51 (72) | 12 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 30 (43) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (28) | 13 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (10)
Dizziness (Nervous system disorders) | 17 (19) | 5 (6)
Headache (Nervous system disorders) | 49 (67) | 33 (39)
Insomnia (Psychiatric disorders) | 24 (24) | 24 (26)
Haematuria (Renal and urinary disorders) | 17 (26) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (45) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (34) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 (39) | 26 (37)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 38 (44) | 8 (9)
Petechiae (Skin and subcutaneous tissue disorders) | 17 (21) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 55 (62) | 24 (32)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (15) | 8 (9)
Hypertension (Vascular disorders) | 26 (34) | 12 (12)
Hypotension (Vascular disorders) | 44 (53) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT02545283/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT02545283/SAP_001.pdf